CLINICAL TRIAL: NCT00928863
Title: Haemorrhagia Postpartum: an Implementation Study on the NVOG Guidelines and MOET Instructions
Acronym: Fluxim
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Rosella Hermens, Dr, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Other Study IDs: 80-82315-98-09003
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Hemorrhage, Postpartum
Keywords: haemorrhagia postpartum; implementation guidelines; maternal morbidity; management of obstetrics and trauma
MeSH Terms: conditions — Postpartum Hemorrhage; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Haemorrhagia post partum: Women with a high risk for haemorrhagia post partum.
  Interventions: Other: implementation aids

INTERVENTIONS:
Other: implementation aids — testing a taylor made strategy for implementation NVOG guideline and MOET instruction in 3 hospitals

SUMMARY:
The objectives of this study is first to asses to what extent the guidelines of the Dutch Society of Obstetrics and Gynaecology (NVOG) and the MOET (Management of Obstetric and Emergencies and Trauma) instructions for haemorrhagia postpartum have been implemented in current care in the Dutch practice. Second to study barriers and facilitators for guideline adherence and to develop and test a tailored implementation strategy, based on these findings.

DETAILED DESCRIPTION:
The most important cause of maternal morbidity in the Netherlands is Haemorrhagia post partum (HPP), with an incidence of 5% containing 10.000 women in the Netherlands a year. Introduction of an evidence-based guideline about HPP by the Dutch society of Obstetrics and Gynaecology (NVOG) and the course Management of Obstetrics Emergencies and Trauma (MOET course) did not lead to a reduction in HPP. This implies the possibility of an incomplete implementation of both the NVOG guideline and MOET-instructions.

To evaluate the implementation of the guideline and MOET instruction in the current care, measurement of the actual care will be performed in a representative sample of 20 hospitals. Before actual care can be measured, quality indicators have to be developed regarding the process, structure and outcome based on the key recommendations from the NVOG guideline on HPP and the MOET instructions. The indicator development will be performed according to the RAND-modified Delphi method .The key recommendations from the NVOG guideline on HPP and the MOET instructions will be extracted and will be tested in two rounds among an independent panel of 12-15. The selected key recommendations will be operationalized in measurable elements. In an observational multi-centre study, actual care will be measured by video monitoring the third stage of delivery and a medical record search among 320 high risk patients for HPP in 20 hospitals. Additional information for indicator adherence will be searched in the medical records of the videotaped patients. In this manner, deviations from the indicators can be outlined. This study will provide us with reliable information about current practice in the Netherlands.

A qualitative study will be performed with the aim to discover factors in detail that are "pro" or "contra" adhering to the developed HPP-indicators by focus group interviews among groups of different involved professionals and experienced patients. Subsequently, to assess the 'prevalence' of the factors mentioned in the focus group interviews, a survey with questionnaires will be performed among all Dutch gynaecologists and midwives. The data will be analyzed to assess the most frequently mentioned barriers and facilitators.

Based on the results of step 1 and 2, a tailored implementation strategy will be developed to increase the adherence to the recommendations. The different implementation elements will be tailored to the barriers and facilitators found and will probably combine interventions directed at professional and organizational level. This strategy will be implemented and evaluated in a feasibility study. The study will be performed in 3 hospitals where the effect of the implementation strategy, the adherence to the developed indicators will be measured. A process evaluation will be performed to study the experiences of the clinicians and patients with this strategy. A cost analysis of the tested implementation strategy will take place.

ELIGIBILITY:
Inclusion Criteria:

* woman with a high risk for haemorrhagia post partum

Exclusion Criteria:

* woman who refuses to participate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women with a high risk for haemorrhagia postpartum delivering in a hospital
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
actual care study: the primary outcome measure is the adherence to the quality indicators (derived from the NVOG guideline on HPP and the MOET instructions). | 1 year
feasibility study: the primary outcome measure regarding effectiveness is the adherence to developed quality indicators. | 1 years
barrier analysis | 1 year
  the primary outcomes in the barrier analysis are the barriers and facilitators among patients and professional regarding adherence to the quality indicators

SECONDARY OUTCOMES:
actual care study: the secondary outcome measure is the outcome (e.g. the incidence of HPP) of care. | 1 year
feasibility study: the secondary outcome measures are the experiences of professionals and patients with the different elements of the implementation strategy and the changed care, and the cost of the tested strategy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rosella Hermens, PhD, Principal Investigator — IQ healthcare, Radboud University Nijmegen Medical Centre
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Woiski M, de Visser S, van Vugt H, Dijkman A, Schuitemaker N, van Meir C, Middeldorp J, Huisjes A, Mol BW, Molkenboer J, Moonen-Delarue D, Oudijk M, van Rheenen-Flach L, Rijnders R, Pernet P, Porath M, de Wit S, Grol R, Scheepers H, Hermens R. Evaluating Adherence to Guideline-Based Quality Indicators for Postpartum Hemorrhage Care in the Netherlands Using Video Analysis. Obstet Gynecol. 2018 Sep;132(3):656-667. doi: 10.1097/AOG.0000000000002781. PMID 30095761
- [Derived] de Visser SM, Woiski MD, Grol RP, Vandenbussche FPHA, Hulscher MEJL, Scheepers HCJ, Hermens RPMG. Development of a tailored strategy to improve postpartum hemorrhage guideline adherence. BMC Pregnancy Childbirth. 2018 Feb 8;18(1):49. doi: 10.1186/s12884-018-1676-6. PMID 29422014
- [Derived] Woiski MD, van Vugt HC, Dijkman A, Grol RP, Marcus A, Middeldorp JM, Mol BW, Mols F, Oudijk MA, Porath M, Scheepers HJ, Hermens RP. From Postpartum Haemorrhage Guideline to Local Protocol: A Study of Protocol Quality. Matern Child Health J. 2016 Oct;20(10):2160-8. doi: 10.1007/s10995-016-2050-9. PMID 27395381
- [Derived] Woiski MD, Belfroid E, Liefers J, Grol RP, Scheepers HC, Hermens RP. Influencing factors for high quality care on postpartum haemorrhage in the Netherlands: patient and professional perspectives. BMC Pregnancy Childbirth. 2015 Oct 23;15:272. doi: 10.1186/s12884-015-0707-9. PMID 26497307
- [Derived] Woiski MD, Hermens RP, Middeldorp JM, Kremer JA, Marcus MA, Wouters MG, Grol RP, Lotgering FK, Scheepers HC. Haemorrhagia post partum; an implementation study on the evidence-based guideline of the Dutch Society of Obstetrics and Gynaecology (NVOG) and the MOET (Managing Obstetric Emergencies and Trauma-course) instructions; the Fluxim study. BMC Pregnancy Childbirth. 2010 Jan 26;10:5. doi: 10.1186/1471-2393-10-5. PMID 20102607